CLINICAL TRIAL: NCT04393363
Title: Early Detection and Prevention of Neuropathy and Cognitive Impairment Following Treatment for Haematological Malignancies (the NOVIT Study)
Brief Title: Early Detection of Neuropathy and Cognitive Impairment Following Treatment for Haematological Malignancies
Acronym: NOVIT1
Status: Active, not recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Marianne Tang Severinsen, Consultant, Head of Research, Ass. Professor, Aalborg University Hospital
Other Study IDs: N-20190068
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: vincristine; bortezomib; lenalidomide; Assessment of nerve fiber excitability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood/plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common, but not well understood complication to treatment with chemotherapy. In this study the investigators will investigate a novel method for early detection of CIPN and compare it to other methods in patients treated for haematological cancers.

DETAILED DESCRIPTION:
Haematological malignancies can be treated with chemotherapy if the patient tolerates the treatment. However, many patients develop complications during treatment including chemotherapy-induced peripheral neuropathy (CIPN) and/or impaired memory. Even though it is a well-known complication, no gold standard for CIPN assessment is known. Besides chemotherapy reduction or cessation, there is so far no sufficient prevention or treatment, therefore early detection and intervention is crucial.

The main purpose of this study is to find a reliable test for chemotherapy-induced peripheral neuropathy (CIPN) in order to predict early signs of CIPN. All included patients has to be scheduled for treatment with vincristine, bortezomib or lenalidomide regardless of haematological malignancy. Neuropathy and cognitive impairment will be tested at baseline (prior to treatment with chemotherapy), before each treatment course, 1 month after treatment and finally 1 year after onset of chemotherapy. CIPN will be examined by different methods: Clinician-based assessment, objective neurophysiological parameters and patient-reported outcome. A novel test using Perception Threshold Tracking (PTT), developed at Aalborg University, is included in the study. The test investigates the nerve excitability in both large and small fiber nerve fibers using two different electrodes. Blood samples will be collected, stored, and analyzed for deficiencies correlated to neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥ 18 years
* Scheduled for treatment with Vincristine (R-CHOP, CHOP, R-CHOEP, CHOEP, R-CVP, CVP or simi-lar), Bortezomib (VCD, MPV, VRD or similar) or Lenalidomide (VRD, len-dex or similar) regardless of type of haematological malignancy
* Not started chemotherapy treatment before enrollment (pretreatment with steroids is allowed)
* Associated to Department of Haematology, Aalborg University Hospital during the project period
* Signed informed consent form
* Able to read and speak Danish

Exclusion Criteria:

* Known vitamin B12 deficiency and treated with either oral or intramuscular vitamin B12 within the last year
* Known neural damage or disease in the neural system (e.g. MS, Guillain-Barre etc.)
* Known severe skin disease
* Pregnancy or breastfeeding
* Inability to understand or comply with instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haematological patients scheduled for (but not started) treatment with vincristine, bortezomib or lenalidomid regardless of type of haematological malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in neuropathy assessed by change in the neurotoxicity (ntx)-subscale of the FACT/GOG-Ntx-13-Score | 0-12 months
  A patient questionnaire with focus on Quality of Life and neuropathy. Range 0-52 with higher score meaning better Quality of Life (less neuropathy). Neuropathy will be defined as a 10 % reduction in the Ntx-score

SECONDARY OUTCOMES:
Change in nerve excitability assessed by Perception Threshold Tracking | 0-12 months
  Assessment of nerve excitability in both large and small fiber nerves measured by two different electrodes.
Change in The National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) | 0-12 months
  A grading scale 1-5 (with 5 as the worst) for neuropathy evaluated by the medical doctor based on the patients' symptoms.
Change in the Total Neuropathy Score-Clinical | 0-12 months
  A score based on clinical evaluation (pin and vibration sensibility, strength and reflexes) and subjective reports from the patient (sensory, motor and autonomic symptoms). The score grades from 0-28 with 28 at worst.
Change in Quality of Life (The total FACT/GOG-Ntx-score) | 0-12 months
  A patient questionnaire with focus on Quality of Life and neuropathy. This part will focus on Quality of Life. Score range from 0-160 with higher score meaning higher Quality of Life
Change in Montreal Cognitive Assessment (MoCA) | 0-12 months
  A quick and easy method to assess mild cognitive disturbance based on following parameters: Awareness, concentration, executive function, memory, abstract thinking, calculating abilities and orientation. The score is 0-30, score > 26 is normal (without cognitive disturbance).
Change in the score for FACT/GOG-cog | 0-12 months
  A patient questionnaire used to assess cognitive function. The score is measured from 0-132 with higher score meaning better Quality of Life
Change in VagusTM Test | 0-12 months
  A measurement for autonomic neuropathy by evaluation of heart rate in different positions
Change in Bioimpendance | 0-12 months
  Measurement of body composition in order to investigate loss of muscle mass, which can influence motor function and imitate or mask motor neuropathy
Change in vitamin B12-level in blood test | 0-12 months
  Measurement of deficiency/functional deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Marianne T Severinsen, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Haematology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maksten EF, Morch CD, Jakobsen LH, Kragholm KH, Blindum PF, Simonsen MR, Ejskjaer N, Dybkaer K, Gregersen H, Madsen J, El-Galaly TC, Severinsen MT. The course of chemotherapy-induced peripheral neuropathy (CIPN) in hematological patients treated with vincristine, bortezomib, or lenalidomide: the NOVIT study. Support Care Cancer. 2025 Feb 26;33(3):225. doi: 10.1007/s00520-025-09282-3. PMID 40011273